CLINICAL TRIAL: NCT02137122
Title: Neuromodulation of Cognition in Older Adults: The Stimulated Brain Study
Brief Title: Neuromodulation of Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201400328-N; 5KL2TR001429 (NIH); 1K01AG050707-01A1 (NIH)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cognitive Training + Active tDCS (Experimental): Participants will undergo up to 10 hours of cognitive training. Cognitive training will involve computerized games that stress elements of cognition. The group will undergo active transcranial direct current stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation
- Cognitive Training + Sham tDCS (Sham Comparator): Participants will undergo up to 10 hours of cognitive training. Cognitive training will involve computerized games that stress elements of cognition. The group will undergo sham transcranial direct current stimulation.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Sham Stimulation — Administer 30 seconds of 2 mA electrical current to the head through saline soaked electrodes.
  Other Names: Soterix 1x1 DC stimulator
  Arms: Cognitive Training + Sham tDCS
Device: Transcranial Direct Current Stimulation — Participants will undergo 20 minutes of 2 mA electrical stimulation to the head through saline soaked electrodes.
  Other Names: Soterix 1x1
  Arms: Cognitive Training + Active tDCS

SUMMARY:
This study will investigate whether transcranial direct current stimulation enhances the effects of cognitive training in healthy older adults.

DETAILED DESCRIPTION:
The current study will investigate methods for enhancing cognitive training effects in healthy older adults by employing a combination of interventions facilitating neural plasticity and optimizing readiness for learning. Adults over the age of 65 represent the fastest growing group in the US population. As such, age-related cognitive decline represents a major concern for public health. Recent research suggests that cognitive training in older adults can improve cognitive performance, with effects lasting up to 10 years. However, these effects are typically limited to the tasks trained, with little transfer to other cognitive abilities or everyday skills. A pilot randomized clinical trial will examine the individual and combined impact of pairing cognitive training with transcranial direct current stimulation (tDCS). tDCS is a method of non-invasive brain stimulation that directly stimulates brain regions involved in active cognitive function and enhances neural plasticity when paired with a training task. We will compare changes in cognitive and brain function resulting from CT and CT combined with tDCS using a comprehensive neurocognitive, clinical, and multimodal neuroimaging assessment of brain structure, function, and metabolic state.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age: 65 to 90 years
* English speaking
* Physically mobile
* working memory function between 0-75th percentile determined by screening results on the POSIT Baseline Cognitive Training computerized tasks.

Exclusion Criteria:

* Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury).
* Evidence of dementia (NACC UDS scores of 1.5 standard deviations below the mean for age, sex and education adjusted norms in a single cognitive domain on the task).
* Past opportunistic brain infection.
* Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality).
* Unstable (e.g., cancer other than basal cell skin) and chronic (e.g, severe diabetes) medical conditions.
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI).
* Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping.
* Certain prescription medications may possibly reduce effects otherwise induced by the tDCS stimulation protocol.
* Hearing or vision deficits that will not allow for standardized cognitive training.
* Left handedness

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Woods, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - McKnight Brain Institute, Gainesville, Florida

REFERENCES:
- [Derived] Nissim NR, O'Shea A, Indahlastari A, Kraft JN, von Mering O, Aksu S, Porges E, Cohen R, Woods AJ. Effects of Transcranial Direct Current Stimulation Paired With Cognitive Training on Functional Connectivity of the Working Memory Network in Older Adults. Front Aging Neurosci. 2019 Dec 16;11:340. doi: 10.3389/fnagi.2019.00340. eCollection 2019. PMID 31998111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Training + Active tDCS | Cognitive Training + Sham tDCS
Started | 15 | 16
Completed | 15 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training + Active tDCS | Cognitive Training + Sham tDCS | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (7.6) | 73.9 (6.7) | 73.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14 | 14 | 28
  African American | 1 | 0 | 1
  Latino | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
NIH toolbox fluid cognition uncorrected standard score [Mean (Standard Deviation); unit: units on a scale] — Scale Name: National Institutes of Health Fluid Cognition Uncorrected Standard Score. Measures constructs of executive function, attention, episodic memory, processing speed and working memory.
  Scores from the flanker test, list sorting working memory test, dimensional change card sort test, pattern comparison processing speed test, and picture sequence memory test are averaged to create the fluid composite.
  Higher values represent better fluid cognition. In this sample, fluid cognition scores ranged from a minimum value of 62 to a maximum value of 111.
  units on a scale | 93.0 (8.6) | 88.9 (12.3) | 90.9 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in NIH Toolbox Fluid Cognition Composite Score
Description: The NIH Toolbox is a battery of neurocognitive tests created by the National Institute on Aging as a comprehensive measure of cognitive function. We used the change from baseline to two week post test in the NIH Toolbox Fluid Cognition Composite Score (FCC) to assess outcome. The uncorrected standard score of the FCC was used. The FCC is derived by averaging the standard scores of the NIH Toolbox Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting, and Pattern Comparison tests and then deriving standard scores based on this new distribution. The uncorrected standard score is on a scale of mean = 100, standard deviation = 15. Higher positive scores mean a greater improvement at the post test. Difference scores ranged from a minimum of -7 to a maximum of 19. FCC scores ranged from a minimum of 73 to a maximum of 112 in this sample. On a population level percentiles are reported from a minimum score of 59 to a maximum of 140, covering 99.3% of the population.
Time Frame: baseline up to two week post test
Population: 1 participant in the Cognitive Training + Sham tDCS group listed in the baseline characteristics section withdrew prior to post test, reducing the number from 16 to 15 in this group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training + Active tDCS | Cognitive Training + Sham tDCS
Number analyzed (Participants) | 15 | 15
units on a scale | 4.7 (7.9) | 6.1 (5.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded between randomization to intervention and three month follow-up.
Arm/Group | Cognitive Training + Active tDCS | Cognitive Training + Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training + Active tDCS (N=15) | Cognitive Training + Sham tDCS (N=16)
Hospitalization (High blood pressure) (Cardiac disorders) | 0 (0) | 1 (1) — Participant was hospitalized due to uncontrolled high blood pressure. Participant reported history of high blood pressure. Hospitalization occurred 89 days post intervention completion and was judged unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02137122/Prot_SAP_000.pdf